CLINICAL TRIAL: NCT04486989
Title: Cardiovascular Conditioning in the Treatment of Vocal Fatigue
Brief Title: Treatment for Teachers With Vocal Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Tennessee State University (Other)
Responsible Party: Principal Investigator, Chayadevie Nanjundeswaran, Associate Professor, East Tennessee State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R15DC017014-01A1 (NIH); 0819.1s-ETSU (Other: East Tennessee State University (ETSU))
Record Dates: First submitted 2020-07-20; First posted 2020-07-27 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Vocal Fatigue; Treatment
MeSH Terms: conditions — Voice Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiovascular Conditioning Protocol (Experimental): Participants will complete a sub maximal cardiovascular training program twice per week for a period of 4 weeks.
  Interventions: Behavioral: Cardiovascular Conditioning Protocol
- Voice Production Exercises (Active Comparator): Participants will complete voice production exercises twice per week for a period of 4 weeks.
  Interventions: Other: Voice Production Exercises

INTERVENTIONS:
Behavioral: Cardiovascular Conditioning Protocol — Participants will be randomized to either one of the treatment arms to receive treatment for a period of 4 weeks.
  Arms: Cardiovascular Conditioning Protocol
Other: Voice Production Exercises — Participants will be randomized to either one of the treatment arms to receive treatment for a period of 4 weeks.
  Arms: Voice Production Exercises

SUMMARY:
Teachers are a population at high risk for voice disorders given their occupational demands. In a teaching career, a common debilitating symptom among all vocal symptoms experienced is - vocal fatigue, impacting teachers' occupational performance and increasing health care costs. It is therefore essential to identify potential treatment options to alleviate the symptom of vocal fatigue. The purpose of this study is to utilize a body-system level cardiovascular training protocol in comparison to traditional voice production training to alleviate the symptoms of vocal fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Female teachers between the ages of 21-60 years Female instructors and college professors between the ages of 21-60 years
* A score of ≥ 15 on factor 1 of the VFI (tiredness and avoidance of voice use) or a score of ≤ 5 on factor 3 of the VFI (improvement of symptoms or lack thereof with rest)
* Sedentary- wherein participants will need to be completing mild intensity cardiovascular exercise less than 150 minutes in less than 5 days per week

Exclusion Criteria:

* Trained athletes
* Trained singers
* Smoking in the past 6months
* Prior history of a vocal fold pathology and current vocal fold pathology

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Changes in Physiologic Cost of Speaking | At baseline, at 4 weeks after treatment
  Physiologic Cost of Speaking is measured as the rate of oxygen consumption at steady state/ rate of speech (wpm) for each of the two reading tasks
Changes in Oxygen Uptake Kinetics | At baseline, at 4 weeks after treatment
  Oxygen Uptake Kinetics is measured as the pattern of oxygen use during each of the two reading tasks
Changes in Post Task Physiological Recovery | At baseline, at 4 weeks after treatment
  Post Task Physiological Recovery is measured as the time, seconds, to reach baseline of oxygen consumption post task (within 0.2ml/kg/min) following each of the reading tasks
Changes in Excess Post Exercise Consumption (EPOC) | At baseline, at 4 weeks after treatment
  EPOC is measured as the magnitude of recovery oxygen consumption, ml/kg/min for each of the reading tasks
Changes in Ratings of Perceived Exertion (RPE) | At baseline, at 4 weeks after treatment
  Borg Scale of Ratings of Perceived Exertion (RPE)- measures the self-report of vocal effort for each of the reading tasks
Changes in Vocal Fatigue Index (VFI) | At baseline, at 4 weeks after treatment
  Vocal Fatigue Index (VFI) is a retrospective scale that measures self-reported symptoms of vocal fatigue
Changes in Global Rating of Vocal Fatigue (VAS 100mm) | At baseline, at 4 weeks after treatment
  Global Rating of Vocal Fatigue (VAS 100mm) measures the ability to sustain voice with no fatigue at the end of a working day

CONTACTS AND LOCATIONS:
Locations (1):
- East Tennessee State University, Johnson City, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/89/NCT04486989/ICF_000.pdf